CLINICAL TRIAL: NCT03849508
Title: Randomized, Double-blind, Controlled Clinical Trial for Comparison of Continuous Phenylephrine Versus Norepinephrine Infusion for Maintenance of Hemodynamic Stability During Cesarean Section Under Spinal Anesthesia
Brief Title: Phenylephrine Versus Norepinephrine for Maintenance of Hemodynamic During Cesarean Section Under Spinal Anesthesia
Acronym: PHENAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHRO-2018-10
Record Dates: First submitted 2019-02-04; First posted 2019-02-21 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Cesarean Section Complications; Spinal Anesthesia
Keywords: cesarean section complications; spinal anesthesia; norepinephrine; maternal hemodynamic and cardiac output
MeSH Terms: interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phenylephrine (Active Comparator): Spinal anesthesia with bupivacaine, sufentanil and morphine will be performed and prophylactic infusion of phenylephrine started at an initial rate of 0,5mcg/kg/ min. The rate will be adjusted according to maternal systolic blood pressure.
  Interventions: Drug: Phenylephrine
- Norepinephrine (Experimental): Spinal anesthesia with bupivacaine, sufentanil and morphine will be performed and prophylactic infusion of norepinephrine tartrate started at an initial rate of 0,1mcg/kg/min. The rate will be adjusted according to maternal systolic blood pressure.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — Drug: Norepinephrine Norepinephrine tartrate variable infusion with a starting rate of 0,1μg/kg/min (equivalent to norepinephrine base of 0.05 μg /Kg/min).
  Other name: Noradrenaline
  Drug: Hyperbaric Bupivacaine will be injected in the subarachnoid space with a dose of 8 to 12 mg adjusted according to height
  Drug: Sufentanil will be injected in the subarachnoid space with a dose of 2,5μg
  Drug: Morphine will be injected in the subarachnoid space with a dose of 100 μg
  Arms: Norepinephrine
Drug: Phenylephrine — Drug: Phenylephrine variable infusion with a starting rate of 0,5μg/kg/min
  Drug: Hyperbaric Bupivacaine will be injected in the subarachnoid space with a dose of 8 to 12 mg adjusted according to height
  Drug: Sufentanil will be injected in the subarachnoid space with a dose of 2,5μg
  Drug: Morphine will be injected in the subarachnoid space with a dose of 100 μg
  Arms: phenylephrine

SUMMARY:
Comparison between prophylactic continuous variable infusion of phenylephrine (starting dose 0,5mcg/kg/min) and norepinephrine tartrate (starting dose 0,1mcg/kg/min) to prevent hypotension and maintain cardiac output under spinal anesthesia during cesarean delivery.

DETAILED DESCRIPTION:
Maternal hypotension is a frequent complication after spinal anesthesia for cesarean delivery. Many vasopressors have been studied and used, but the perfect vasopressor is yet to be found. Phenylephrine is the most common used in obstetric anesthesia but its cardiac depressant activity, being an only alpha-adrenergic agonistic, is linked to frequent side effects such as bradycardia and decreased cardiac output.

Norepinephrine is a vasopressor characterized by both alpha and minor beta-adrenergic agonistic activity, it has then a minimal cardiac depressant activity. Hence it would provide a better stability of hemodynamic and cardiac output, and appears as a better alternative to phenylephrine.

In this study, the investigators will compare prophylactic continuous variable infusion of both vasopressors. Phenylephrine started at the dose of 0,5mcg/kg/min and Norepinephrine tartrate started at the dose of 0,1mcg/kg/min. The doses will be adjusted according to maternal systolic blood pressure in order to prevent hypotension (defined by a systolic blood pressure under 80% of baseline).

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy higher than 36 weeks of amenorrhea
* Scheduled or semi-urgent (interval between decision and delivery by cesarean section higher than 12hours) cesarean section under spinal anesthesia

Exclusion Criteria:

* Extreme height (less than 140cm; higher than 180cm)
* Weight less than 50kg
* Weight higher than 120kg
* Cardiovascular disease with use of cardiac medication (including antihypertensive drug)
* Active neurological disease
* Anti-hypertension treatment.
* High blood pressure or severe pre-eclampsia
* American Society of Anesthesiologists physical status class higher than 3
* Placenta accrete/percreta
* Cesarean section scheduled under general anesthesia
* Contraindications to spinal anesthesia
* Minor (age less than 18 years old)
* Guardianship/ curatorship
* Anemia less than or equal to 8 g/dl
* Allergy to any study medication
* Simultaneous participation in another study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 124 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Cardiac output maintenance (measured in L/min by bioreactance). | 5 minutes before the induction of spinal anesthesia until umbilical cord clamping.
  Cardiac output values were analyses at eight points
  * Baseline measurement: patient placed in the supine position with the table tilted 10° left, before spinal anesthesia
  * Seven measurements at regular intervals: first measurement just after administration of spinal anesthesia in supine position with the table tilted 10° left and last measurement at umbilical cord clamping.

SECONDARY OUTCOMES:
Heart rate | From induction of spinal anesthesia until weaning of vasopressor
  number of heart beats per minute
Systolic blood pressure | From induction of spinal anesthesia until weaning of vasopressor
  Systolic blood pressure measured in mmHg
Mean blood pressure | From induction of spinal anesthesia until weaning of vasopressor
  Mean blood pressure measured in mmHg
Duration of bradycardia | From induction of spinal anesthesia until weaning of vasopressor]
  Cumulative time in minutes with heart rate less than 60 beats/min
Duration of hypotension with Mean blood pressure less than 65mmHg | after applying spinal anesthesia until weaning of vasopressor
  Cumulative time in minutes
Duration of hypotension with Systolic Blood Pressure less than 80mmHg | after applying spinal anesthesia until weaning of vasopressor
  Cumulative time in minutes
Duration of hypertension | after applying spinal anesthesia until weaning of vasopressor
  Cumulative time in minutes with Systolic Blood Pressure more than 140mmHg
Cardiac Output | after applying spinal anesthesia until weaning of vasopressor
  Measured in L/min
Stroke Volume | after applying spinal anesthesia until weaning of vasopressor
  Measured in ml/beat
Total Peripheral Resistance | after applying spinal anesthesia until weaning of vasopressor
  Measured in dynes.sec.cm-5
Maximum flow rate of study drug given | after applying spinal anesthesia until weaning of vasopressor
  Measured in mcg/hour
Total dose of study drug consumed | after applying spinal anesthesia until weaning of vasopressor
  Total dose of study drug given from induction of spinal anesthesia to delivery of the fetus
Total Rescue Bolus Dose of atropine to maintain Systolic Blood Pressure | after applying spinal anesthesia until weaning of vasopressor
  Total dose of atropine administered (mg)
Total Rescue Bolus Dose of ephedrine or other vasopressor to maintain Systolic Blood Pressure | after applying spinal anesthesia until weaning of vasopressor
  Total dose of ephedrine or other vasopressor administered (mg)
Incidence of nausea or vomiting | after applying spinal anesthesia until weaning of vasopressor
  The percentage of patients with nausea or vomiting (at least one episode)
Incidence of dizziness or malaise | after applying spinal anesthesia until weaning of vasopressor
  The percentage of patients with dizziness or malaise (at least one episode)
Maternal blood glucose concentration | at peripheral intravenous line placement
  concentration measured in mmol/l
Maternal blood glucose concentration | at umbilical cord clamping
  concentration measured in mmol/l
APGAR score | 1 minute after delivery
  APGAR score of the fetus ranging from 0 to 10
APGAR score | 3 minutes after delivery
  APGAR score of the fetus ranging from 0 to 10
APGAR score | 5 minutes after delivery
  APGAR score of the fetus ranging from 0 to 10
APGAR score | 10 minutes after delivery
  APGAR score of the fetus ranging from 0 to 10
Umbilical arterial potential hydrogen | At time of birth
  potential hydrogen in the blood sample obtained from umbilical artery scaled from 1 to 14
Fetal lactates | At time of birth
  from umbilical artery blood sample, measured in mmol/l
Umbilical arterial partial pressure of carbon dioxide | At time of birth
  in the blood sample obtained from umbilical artery measured in mmHg
Umbilical arterial partial pressure of oxygen | At time of birth
  in the blood sample obtained from umbilical artery measured in mmHg
Umbilical arterial base excess | At time of birth
  in the blood sample obtained from umbilical artery measured in mmol/L
Fetal blood glucose concentration at birth | At time of birth
  from umbilical artery blood sample, measured in mmol/l
Neonatal blood glucose concentration | at 1 hour after birth
  Capillary blood glucose is measured in mmol/l
Uterine and umbilical arteries Doppler with measurement of the pulsatility | 5 minutes before realization of spinal anesthesia
  pulsatility index of Gosling (peak systolic velocity - end diastolic velocity /mean velocity)
Uterine and umbilical arteries Doppler with measurement of the pulsatility | 5 minutes after induction of spinal anesthesia
  pulsatility index of Gosling (peak systolic velocity - end diastolic velocity /mean velocity)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BELIN, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- Regional Hospital Center of ORLEANS, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mercier FJ, Auge M, Hoffmann C, Fischer C, Le Gouez A. Maternal hypotension during spinal anesthesia for caesarean delivery. Minerva Anestesiol. 2013 Jan;79(1):62-73. Epub 2012 Nov 18. PMID 23135692
- [Background] Langesaeter E, Dyer RA. Maternal haemodynamic changes during spinal anaesthesia for caesarean section. Curr Opin Anaesthesiol. 2011 Jun;24(3):242-8. doi: 10.1097/ACO.0b013e32834588c5. PMID 21415724
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Chooi C, Cox JJ, Lumb RS, Middleton P, Chemali M, Emmett RS, Simmons SW, Cyna AM. Techniques for preventing hypotension during spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2017 Aug 4;8(8):CD002251. doi: 10.1002/14651858.CD002251.pub3. PMID 28976555
- [Background] Stewart A, Fernando R, McDonald S, Hignett R, Jones T, Columb M. The dose-dependent effects of phenylephrine for elective cesarean delivery under spinal anesthesia. Anesth Analg. 2010 Nov;111(5):1230-7. doi: 10.1213/ANE.0b013e3181f2eae1. Epub 2010 Sep 14. PMID 20841418
- [Background] Ngan Kee WD. The use of vasopressors during spinal anaesthesia for caesarean section. Curr Opin Anaesthesiol. 2017 Jun;30(3):319-325. doi: 10.1097/ACO.0000000000000453. PMID 28277383
- [Background] Vallejo MC, Attaallah AF, Elzamzamy OM, Cifarelli DT, Phelps AL, Hobbs GR, Shapiro RE, Ranganathan P. An open-label randomized controlled clinical trial for comparison of continuous phenylephrine versus norepinephrine infusion in prevention of spinal hypotension during cesarean delivery. Int J Obstet Anesth. 2017 Feb;29:18-25. doi: 10.1016/j.ijoa.2016.08.005. Epub 2016 Aug 28. PMID 27720613
- [Background] Ngan Kee WD, Lee SWY, Ng FF, Khaw KS. Prophylactic Norepinephrine Infusion for Preventing Hypotension During Spinal Anesthesia for Cesarean Delivery. Anesth Analg. 2018 Jun;126(6):1989-1994. doi: 10.1213/ANE.0000000000002243. PMID 28678073
- [Background] McLaughlin K, Wright SP, Kingdom JCP, Parker JD. Clinical Validation of Non-Invasive Cardiac Output Monitoring in Healthy Pregnant Women. J Obstet Gynaecol Can. 2017 Nov;39(11):1008-1014. doi: 10.1016/j.jogc.2017.02.015. Epub 2017 Jul 18. PMID 28733057
- [Derived] Belin O, Casteres C, Alouini S, Le Pape M, Dupont A, Boulain T. Manually Controlled, Continuous Infusion of Phenylephrine or Norepinephrine for Maintenance of Blood Pressure and Cardiac Output During Spinal Anesthesia for Cesarean Delivery: A Double-Blinded Randomized Study. Anesth Analg. 2023 Mar 1;136(3):540-550. doi: 10.1213/ANE.0000000000006244. Epub 2022 Oct 24. PMID 36279409